CLINICAL TRIAL: NCT02817633
Title: A Phase 1 Dose Escalation and Cohort Expansion Study of TSR-022, an Anti-TIM-3 Monoclonal Antibody, in Patients With Advanced Solid Tumors (AMBER)
Brief Title: A Study of TSR-022 in Participants With Advanced Solid Tumors (AMBER)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 213348; 2018-002143-29 (EudraCT Number); NCT06322693 (obsolete NCT alias)
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Neoplasms
Keywords: TSR-022; Nivolumab; Advanced solid tumors; Metastatic solid tumors; Immunotherapy; Colorectal cancer; Non-small cell lung cancer; Melanoma; TSR-033; TSR-042; Hepatocellular carcinoma cancer; Docetaxel
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — Nivolumab; dostarlimab; TSR-033; Docetaxel; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a multi-center, open-label, first-in-human Phase 1 study.
Masking Description: Click here to enter text.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Part 1a: TSR-022 monotherapy (Experimental)
  Interventions: Drug: TSR-022
- Part 1b: TSR-022 in combination with nivolumab (Experimental)
  Interventions: Drug: TSR-022; Drug: Nivolumab
- Part 1c: TSR-022 in combination with TSR-042 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042
- Part 1d: TSR-022 in combination with TSR-042 and TSR-033 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042; Drug: TSR-033
- Part 1e: TSR-022 with TSR-042 (not previously treated with anti-programmed death ligand [PD-{L}]1) (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042
- Part 1f: TSR-022 in combination with TSR-042 and Docetaxel (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042; Drug: Docetaxel
- Part 1g: TSR-022 in combination with TSR-042, pemetrexed, and cisplatin (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042; Drug: Pemetrexed; Drug: Cisplatin
- Part 1h: TSR-022 in combination with TSR-042, pemetrexed, and carboplatin (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042; Drug: Pemetrexed; Drug: Carboplatin
- Part 2: Cohort A Melanoma-TSR-022 as monotherapy (Experimental)
  Interventions: Drug: TSR-022
- Part 2: Cohort A Melanoma-TSR-022 with TSR-042 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042
- Part 2:Cohort B Non-small cell lung cancer-TSR-022-monotherapy (Experimental)
  Interventions: Drug: TSR-022
- Part 2:Cohort B Non-small cell lung cancer-TSR-022 with TSR-042 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042
- Part 2:Cohort C Colorectal cancer-TSR-022 as monotherapy (Experimental)
  Interventions: Drug: TSR-022
- Part 2:Cohort C Colorectal cancer-TSR-022 with TSR-042 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042
- Part 2: Cohort D-TIM-3 selected non-small cell lung cancer (NSCLC)-TSR-022 with TSR-042 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042
- Part 2: Cohort E-Non-small cell lung cancer-TSR-022 with docetaxel (Experimental)
  Interventions: Drug: TSR-022; Drug: Docetaxel
- Part 2: Cohort F- Hepatocellular carcinoma (HCC)-TSR-022 with TSR-042 (Experimental)
  Interventions: Drug: TSR-022; Drug: TSR-042

INTERVENTIONS:
Drug: TSR-022 — TSR-022 will be administered.
Drug: Nivolumab — Nivolumab will be administered.
  Arms: Part 1b: TSR-022 in combination with nivolumab
Drug: TSR-042 — TSR-042 will be administered.
  Arms: Part 1c: TSR-022 in combination with TSR-042; Part 1d: TSR-022 in combination with TSR-042 and TSR-033; Part 1e: TSR-022 with TSR-042 (not previously treated with anti-programmed death ligand [PD-{L}]1); Part 1f: TSR-022 in combination with TSR-042 and Docetaxel; Part 1g: TSR-022 in combination with TSR-042, pemetrexed, and cisplatin; Part 1h: TSR-022 in combination with TSR-042, pemetrexed, and carboplatin; Part 2: Cohort A Melanoma-TSR-022 with TSR-042; Part 2: Cohort D-TIM-3 selected non-small cell lung cancer (NSCLC)-TSR-022 with TSR-042; Part 2: Cohort F- Hepatocellular carcinoma (HCC)-TSR-022 with TSR-042; Part 2:Cohort B Non-small cell lung cancer-TSR-022 with TSR-042; Part 2:Cohort C Colorectal cancer-TSR-022 with TSR-042
Drug: TSR-033 — TSR-033 will be administered.
  Arms: Part 1d: TSR-022 in combination with TSR-042 and TSR-033
Drug: Docetaxel — Docetaxel will be administered.
  Arms: Part 1f: TSR-022 in combination with TSR-042 and Docetaxel; Part 2: Cohort E-Non-small cell lung cancer-TSR-022 with docetaxel
Drug: Pemetrexed — Pemetrexed will be administered.
  Arms: Part 1g: TSR-022 in combination with TSR-042, pemetrexed, and cisplatin; Part 1h: TSR-022 in combination with TSR-042, pemetrexed, and carboplatin
Drug: Cisplatin — Cisplatin will be administered.
  Arms: Part 1g: TSR-022 in combination with TSR-042, pemetrexed, and cisplatin
Drug: Carboplatin — Carboplatin will be administered.
  Arms: Part 1h: TSR-022 in combination with TSR-042, pemetrexed, and carboplatin

SUMMARY:
This is a first-in-human study evaluating the anti-T cell immunoglobulin and mucin containing protein-3 (TIM-3) antibody TSR-022. The study will be conducted in 2 parts with Part 1 consisting of dose escalation and Part 2 dose expansion. Part 1 will determine the recommended Phase 2 dose (RP2D) of TSR-022 and Part 2 will evaluate the antitumor activity of TSR-022 in combination with TSR-042 or docetaxel and as monotherapy.

ELIGIBILITY:
Inclusion Criteria

* Participant is at least 18 years of age.
* Female participants of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the date of the first dose of study medication or be of non-childbearing potential.
* Participant has an ECOG performance status of less than or equal to (<=)1.
* Participant has adequate organ function.

Inclusion Criteria for Participants in Part 1 and Part 2 Cohorts A, B, and C:

* Participant with advanced or metastatic solid tumor who meets the requirements for the part of the study/cohort he/she will participate in, as follows:
* Part 2: Histologically proven advanced (unresectable) or metastatic solid tumor that is measurable by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST version 1.1 criteria Inclusion Criteria for Participants in Part 2 Cohort D
* Participants with advanced or metastatic non-small cell lung carcinoma (NSCLC) that is measurable by CT or MRI per RECIST version 1.1 criteria and meet the following criteria:
* NSCLC histology includes squamous or non-squamous cell carcinoma.
* Participants have received no more than 2 prior lines of therapy, which must include a platinum-based chemotherapy (for example [e.g.], cisplatin, carboplatin) and an anti- programmed death-ligand 1 (PD-L1) antibody.
* Participants must have documented radiographic progression by RECIST version 1.1 criteria on prior anti-programmed cell death protein (PD-1) or anti-PD-L1 therapy.
* Biopsies -All participants enrolled must undergo a biopsy prior to study entry, and the biopsy tissue must be submitted to the central laboratory for all participants in order to determine T-cell immunoglobulin and mucin-domain containing-3 (TIM-3) expression level prior to first dose. If a participant has had a biopsy prior to entering the 35-day screening period and within approximately 12 weeks of study treatment, that biopsy may be accepted as the Baseline fresh biopsy.

Inclusion Criteria for Participants in Part 2 Cohort E

* Participant is greater than or equal to (>=)18 years old, is able to understand the study procedures, and agrees to participate in the study by providing written informed consent which includes compliance with the requirements and restrictions listed in the Informed consent form (ICF) and protocol.
* Participant has histologically or cytologically proven advanced or metastatic NSCLC, and only squamous or non-squamous cell carcinoma.
* Participant has received no more than 2 prior lines of therapy for advanced or metastatic disease, which must only include a platinum-based (eg, cisplatin, carboplatin) doublet chemotherapy regimen and an anti-PD-1 or anti-PD-L1 antibody (no other biologic agents alone or in combination; novel combinations are not allowed). Participants previously treated with targeted therapies, including angiogenesis inhibitors (eg, bevacizumab, ramucirumab, lenvatinib), are not eligible.
* Participant has measurable disease, that is, presenting with at least 1 measurable lesion per RECIST v1.1 as determined by the local site Investigator/radiology assessment. Target lesions situated in a previously irradiated area are considered measurable if disease progression has been demonstrated in such lesions and if there are other target lesions. If there is only 1 target lesion that was previously irradiated, the participant is not eligible.
* Participant has documented radiological disease progression on prior platinum-based chemotherapy and on prior anti-PD-1 or anti-PD-L1 therapy according to RECIST v1.1.
* Participant agrees to submit an archival formalin fixed paraffin embedded (FFPE) tumor tissue specimen that was collected on or after diagnosis of metastatic disease from location(s) not irradiated prior to biopsy. Both tissue block and freshly cut slides are acceptable. If archival tissue is not available, the participant must undergo biopsy prior to study entry.
* Participant has an ECOG performance status score of 0 or 1.
* Participant has a life expectancy of at least 3 months and is anticipated to be able to complete 4 cycles of docetaxel treatment.
* Participant has adequate organ function as defined in the protocol
* Contraceptive use by male and female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Inclusion Criteria for Participants in Part 2 Cohort F

* Histologically confirmed locally advanced or metastatic and/or unresectable Hepatocellcular Carcinoma (HCC)

  * Barcelona Clinic Liver Cancer Stage B or C
  * Cirrhosis grade of Child-Pugh Class A
* No prior systemic therapy for HCC
* Documented HBV testing at screening, including hepatitis B surface antigen (HBsAg), hepatitis B surface antibody (HBsAB) and hepatitis B core antibody (HBcAb). Participants with a positive HBsAg will require negative hepatitis B virus (HBV) DNA testing at screening.

  * Participants with chronic HBV infection (HBsAg +) are required to be receiving effective antiviral therapy (i.e., with Tenofovir or Entecavir) for at least 14 days with willingness to continue for the length of the study and have HBV deoxyribonucleic acid (DNA) less than 100 International Units Per Milliliter (IU/mL) within 28 days prior to initiation of study treatment.
  * Participants with chronic HBV infection (HBsAg+) require documented Hepatitis D virus (HDV) antibody testing conducted at screening. If HDV antibody is positive, then HDV ribonucleic acid (RNA) must be negative to participate.
  * Participants with a negative HBsAg and positive HBcAb result are eligible only if HBV DNA is negative (Past HBV participants).
* Documented hepatitis C virus (HCV) antibody testing conducted at screening. If HCV antibody is positive, then HCV RNA must be negative. Participants with recently treated HCV prior to study start must be greater than (>)12 weeks from final HCV treatment.
* Must have measurable disease, defined as at least one tumor lesion that can be accurately measured according to RECIST v1.1
* Participant agrees to submit an archival FFPE tumor tissue specimen that was collected on or after diagnosis of metastatic disease from location(s) not irradiated prior to biopsy. Both tissue block and freshly cut slides are acceptable. If archival tissue is not available, the participant must undergo biopsy prior to study entry.

  • Participants are also encouraged, but not required, to have a fresh tumor tissue biopsy of a primary or metastatic tumor prior to dosing (samples will be used to enable biomarker analysis).
* International normalized ratio (INR) or prothrombin time (PT) <= 2× upper limit of normal (ULN) unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin (PTT) is within therapeutic range of intended use of anticoagulants. Activated partial thromboplastin time (aPTT) <=2×ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Negative human immunodeficiency virus (HIV) test at screening The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

Exclusion criteria:

* History of Grade greater than or equal to (>=)3 immune-related AE with prior immunotherapy, with the exception of non-clinically significant lab abnormalities.
* Participant has known uncontrolled central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Participant has a known additional malignancy that progressed or required active treatment within the last 2 years. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the Medical Monitor.
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active infection requiring systemic therapy.
* Participant is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the Screening Visit through 150 days after the last dose of study treatment.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.

Exclusion Criteria for Participants in Part 2 Cohort D

* A participant with negative (as determined by Central Testing Lab) or unevaluable TIM-3 expression from tissue obtained prior to study entry will not be eligible for the study.
* Participant has received prior therapy as defined below:
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agent that resulted in permanent discontinuation due to an AE.
* Prior treatment with an anti-lymphocyte activation gene (LAG)-3 or anti-TIM-3.
* Radiologic or clinical progression <= 8 weeks after initiation of prior anti-PD-1 or anti-PD-L1 antibody.
* Participants with known epidermal growth factor receptor (EGFR) mutation, anaplastic lymphoma kinase (ALK) translocation, or receptor tyrosine kinase (ROS1) mutation.
* Participant has received a vaccine other than a vaccine against severe acute respiratory syndrome (SARS)-coronavirus 2 (CoV-2) infection ("Coronavirus Disease 2019" [COVID-19]) within 7 days of planned start of study therapy. The use of all COVID-19 vaccines is allowed, with the exception of COVID-19 vaccines using the recombinant adenoviral vector platform within 30 days of planned start of study therapy. If a COVID-19 vaccine using this platform is to be administered within 30 days of planned start of study therapy, this must first be discussed with and approved by the Sponsor's Medical Monitor.

Exclusion Criteria for Participants in Part 2 Cohort E

* Participant has been previously treated with an anti PD 1, anti PD L1, or anti PD L2 agent that resulted in permanent discontinuation due to an AE
* Participant has been previously treated with an anti TIM-3 or anti cytotoxic T lymphocyte-associated protein 4 (CTLA 4) agent or docetaxel.
* Participant has a documented sensitizing EGFR, ALK, or ROS-1 mutation. Participants whose tumors have not been tested for these driver mutations and therefore who have unknown driver mutation status are not eligible. Participants with squamous histology do not need to be tested for these driver mutations.
* Participant had radiological or clinical disease progression (that is [ie,] worsening performance status, clinical symptoms, and laboratory data) <=8 weeks after initiation of prior anti PD 1 or anti-PD-L1 antibody. The clinical disease progression should have been confirmed by a subsequent radiological scan.
* Participant has received radiation to the lung that is >30 Gray (Gy) within 6 months prior to the first dose of study treatment.
* Participant has completed palliative radiotherapy within 7 days prior to the first dose of study treatment.
* Participant has an additional malignancy or a history of prior malignancy, with the exception of adequately treated basal or squamous skin cancer, cervical carcinoma in situ, or bladder carcinoma in situ without evidence of disease, or had a malignancy treated with curative intent and with no evidence of disease recurrence for 5 years since the initiation of that therapy.
* Participant has known new or progressive brain metastases and/or leptomeningeal metastases. Participants who have received prior therapy for their brain metastases and have radiologically stable central nervous system disease may participate, provided they are neurologically stable for at least 4 weeks before study entry and are off corticosteroids within 3 days prior to the first dose of study treatment.
* Participant has tested positive for the following at Screening or within 3 months before the first dose of study treatment:
* Presence of hepatitis B surface antigen.
* Presence of hepatitis C antibody in the absence of an Ribonucleic acid (RNA) test for hepatitis C virus.
* Participant has known human immunodeficiency virus (HIV) (positive for HIV 1 or HIV 2 antibodies).
* Participant has active autoimmune disease that required systemic treatment in the past 2 years, is immunocompromised in the opinion of the Investigator, or is receiving systemic immunosuppressive treatment. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy of prednisone, or equivalent, for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Participant has received systemic steroid therapy within 3 days prior to the first dose of the study treatment or is receiving any other form of immunosuppressive medication. Replacement therapy is not considered a form of systemic therapy. Use of inhaled corticosteroids, local steroid injection, or steroid eye drops is allowed.
* Participant has current interstitial lung disease, current pneumonitis, or a history of pneumonitis that required the use of glucocorticoids to assist with management. Lymphangitic spread of the NSCLC is not exclusionary.
* Participant does not meet requirements per local prescribing guidelines for receiving treatment with docetaxel, including severe hypersensitivity reactions to drugs formulated with polysorbate 80.
* Participant has received prior anticancer therapy (chemotherapy, targeted therapies, radiotherapy, or immunotherapy) within 21 days, or less than 5 times the half life of the most recent therapy prior to study Day 1, whichever is shorter.

Exclusion Criteria for Participants in Part 2 Cohort F

* Known fibrolamellar HCC, sarcomatoid HCC or mixed cholangiocarcinoma and HCC
* Participant must not have had major surgery <= 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects
* Participants must not have received investigational therapy <= 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating protocol therapy.
* Active or untreated central nervous system (CNS) and leptomeningeal metastases
* Prior therapy with any medication targeting PD-1, PD-L1, or TIM-3
* Participant must not have a known hypersensitivity to TSR-042 and TSR-022 components or excipients.
* Participants with active malignancy (other than HCC) or a prior malignancy within the past 2 years are excluded. Participants with completely resected cutaneous melanoma (early stage), basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and localized prostate cancer are eligible
* Participant must not have serious, uncontrolled medical disorder, or nonmalignant systemic disease as determined by the treating physician. Examples include, but are not limited to uncontrolled ventricular arrhythmia, uncontrolled major seizure disorder, unstable spinal cord compression, or superior vena cava syndrome.
* Has a history or evidence of cardiac abnormalities within the 6 months prior to enrollment, including:

  * Serious, uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities including second-degree (Type II) or third-degree atrioventricular (AV) block.
  * Cardiomyopathy, myocarditis, myocardial infarction, acute coronary syndromes (including angina pectoris), coronary angioplasty, stenting, or bypass grafting.
  * Congestive heart failure [New York Heart Association (NYHA) Class III or IV]
  * Symptomatic pericarditis
* Known history of HIV infection
* Active tuberculosis infection or other microbial infection or any active systemic infection requiring parenteral antibiotic therapy. All prior infections must have resolved following optimal therapy.
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years (. i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of idiopathic pulmonary fibrosis, interstitial lung disease, bronchial asthma, organizing pneumonia, bronchiolitis obliterans, drug-induced pneumonitis, or idiopathic pneumonitis
* History of organ transplantation including allogeneic bone marrow transplantation
* Participant has a diagnosis of immunodeficiency or has been receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy.
* Participant has received a live vaccine within 7 days of initiating protocol therapy. Seasonal flu vaccines that do not contain live virus and COVID 19 vaccines are permitted.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant, lactating, breastfeeding, or intending to become pregnant during the study and for 150 days after the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 (a): Number of participants achieving dose limiting toxicity (DLTs) | Up to 28 days
Part 1 (b,c,d): Number of participants achieving dose limiting toxicity (DLTs) | Up to 42 days
Part 1 (f,g,h): Number of participants achieving dose limiting toxicity (DLTs) | Up to 21 days
Part 1: Number of participants with adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation, treatment emergent adverse events (TEAEs), TEAEs leading to death and immune-related adverse events (irAEs) | Up to 2 years
Part 1: Number of participants with clinically significant changes in laboratory parameters, vital signs, electrocardiogram (ECG) findings, Eastern Cooperative Oncology Group (ECOG) status, physical examination and use of concomitant medications | Up to 2 years
Part 1 (e) and Part 2: Overall Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 | Up to 2 years

SECONDARY OUTCOMES:
Part 1 (a, b, c, d, f, g, h): ORR by RECIST v 1.1 | Up to 2 years
Part 2 (A, B, C, D): ORR by Immune related RECIST (irRECIST) | Up to 2 years
Part 2: Duration of response (DOR) by RECIST v 1.1 | Up to 2 years
Part 2 (A, B, C, D): DOR by irRECIST | Up to 2 years
Parts 1 and 2: Disease control rate (DCR) by RECIST v 1.1 | Up to 2 years
Part 2 (A, B, C, D): DCR by irRECIST | Up to 2 years
Part 2: Progression-free survival (PFS) by RECIST v 1.1 | Up to 2 years
Part 2 (A, B, C, D): PFS by irRECIST | Up to 2 years
Parts 1 and 2 (A, B, C, D, E, F): Serum concentration of TSR-022 | Up to 2 years
Part 1d: Serum concentration of TSR-033 | Up to 2 years
Part 1 (c, d, e, f, g, h): Serum concentration of TSR-042 | Up to 2 years
Part 2 (A, B, C, D, F): Serum concentration of TSR-042 | Up to 2 years
Part 2: Overall survival (OS) | Up to 2 years
Part 1a: Minimum plasma concentration (Cmin) of TSR-022 as monotherapy | Up to 2 years
Part 1b: Cmin of TSR-022 in combination with nivolumab | Up to 2 years
Part 1c: Cmin of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1d: Cmin of TSR-022 in combination with TSR-042 and TSR-033 | Up to 2 years
Part 2F: Cmin of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1a: Area under the concentration × time curve from time 0 to infinity AUC (0-inf) of TSR-022 as monotherapy | Up to 2 years
Part 1b: AUC (0-inf) of TSR-022 in combination with nivolumab | Up to 2 years
Part 1c: AUC (0-inf) of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1d: AUC (0-inf) of TSR-022 in combination with TSR-042 and TSR-033 | Up to 2 years
Part 2F: AUC (0-inf) of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1a: Area under the concentration time curve from time 0 to last assessment (AUC 0-last) of TSR-022 as monotherapy | Up to 2 years
Part 1b: AUC (0-last) of TSR-022 in combination with nivolumab | Up to 2 years
Part 1c: AUC (0-last) of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1d: AUC (0-last) of TSR-022 in combination with TSR-042 and TSR-033 | Up to 2 years
Part 2F: AUC (0-last) of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1a: Terminal half life (t 1/2) of TSR-022 as monotherapy | Up to 2 years
Part 1b: t1/2 of TSR-022 and in combination with nivolumab | Up to 2 years
Part 1c: t1/2 of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1d: t1/2 of TSR-022 in combination with TSR-042 and TSR-033 | Up to 2 years
Part 2F: t1/2 of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1a: Area under the concentration × time curve during the dosing interval (AUCtau) of TSR-022 as monotherapy | Up to 2 years
Part 1b: AUCtau of TSR-022 and in combination with nivolumab | Up to 2 years
Part 1c: AUCtau of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1d: AUCtau of TSR-022 in combination with TSR-042 and TSR-033 | Up to 2 years
Part 2F: AUCtau of TSR-022 in combination with TSR-042 | Up to 2 years
Part 1: Number of participants with anti-drug antibodies (ADAs) to TSR-022 | Up to 2 years
Part 2 (A, B, C, D, E, F): Number of participants with ADA to anti-TSR-022 | Up to 2 years
Part 1 (c, d, e, f, g, h): Number of participants with ADA to TSR-042 | Up to 2 years
Part 2 (A, B, C, D, F): Number of Participants with ADA to TSR-042 | Up to 2 years
Part 1d: Number of participants with ADA to TSR-033 | Up to 2 years
Part 2F: Number of participants with AEs, SAEs, AEs leading to discontinuation, TEAEs, TEAEs leading to death | Up to 2 years
Part 2F: Percent change from Baseline in Alpha-fetoprotein (AFP) | Baseline, and up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (74):
- United States (59):
  - GSK Investigational Site, Goodyear, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Encinitas, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Marcos, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Arlington Heights, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Niles, Illinois
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Pikeville, Kentucky
  - GSK Investigational Site, Wheaton, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Florissant, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hackensack, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Vancouver, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Kennewick, Washington
  - GSK Investigational Site, Puyallup, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Madison, Wisconsin
- South Korea (2):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
- Spain (13):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, L'Hospitalet de Llobrega
  - GSK Investigational Site, Las Palmas de Gran Canar
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No